CLINICAL TRIAL: NCT00847730
Title: A Single Arm, Prospective Clinical Trial Evaluating the Ease of Use of a VAC GranuFoam Bridge Dressing on Diabetic Foot Ulcers Receiving VAC Negative Pressure Therapy
Brief Title: Evaluating the Ease of Use of a VAC GranuFoam Bridge Dressing on Diabetic Foot Ulcers Receiving VAC Negative Pressure Wound Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VACDrsg 2008-37
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Ulcers
Keywords: Ease of dressing application, dressing conformability and ease of dressing removal on diabetic foot ulcers using the ActiVAC therapy
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VAC GranuFoam Bridge Dressing (Experimental): This is a medical device foam dressing allowing placement away from wound site. It is designed to simplify the bridging application. It is used in combination with the V.A.C. Negative Pressure Wound Therapy System. For each subject, the dressing was applied in compliance with the IFU for 48-72 hours.
  Interventions: Device: V.A.C. Negative Pressure Wound Therapy System

INTERVENTIONS:
Device: V.A.C. Negative Pressure Wound Therapy System — This is a non-invasive wound treatment system that uses controlled, localized negative pressure to create an environment that promotes wound healing in chronic and acute wounds

SUMMARY:
The study is aimed at evaluating the clinician's perceived ease of using the V.A.C. GranuForm bride dressing and the patients perceived level of comfort during the dressing wear.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the ease of use of the V.A.C® GranuFoam™ Bridge dressing on Diabetic Foot Ulcers under ActiV.A.C® negative pressure wound therapy for a period of 48-72 hrs (+6hrs). Ease of use will be determined based on the feedback on the following characteristics 1) Ease of dressing application 2) Ease of dressing removal and 3) Ease of dressing conformability. Additionally patient feedback on comfort during wear will also be collected. Patients currently prescribed to V.A.C.® Therapy will be enrolled in the trial.

ELIGIBILITY:
Inclusion Criteria

1. Male or Female subjects must be ≥ 18 years of age
2. Subject is willing and able to provide written informed consent and comply with protocol required procedures
3. Subject has a calcaneal, dorsal or plantar diabetic foot ulcer no greater than a Grade 2 on the Wagner Grading System for which ActiV.A.C.® Therapy has been prescribed and requires off loading of the SensaT.R.A.C. PadTM
4. Subject has a foot ulcer that is ≥ 1.5cm2 but no greater than 84 cm2
5. Female subject that is willing to use an effective method of contraception for the duration of the study, is permanently sterilized, or post-menopausal as defined by cessation of menses for at least twelve (12) months prior to enrollment. Acceptable means of contraception is defined as use of Birth control pills, Depo Provera® , Norplant® , IUD (intrauterine device), Diaphragm with spermicide, Condom with spermicide

Exclusion Criteria

1. Subject's wound measures > 84 cm2
2. Presence of untreated cellulitis
3. Presence of untreated or refractory osteomyelitis (including untreated necrotic bone, non-viable tissue and infected bone)
4. History of radiation to the wound area
5. History of thermal injury in the wound area
6. Known hypersensitivity to any disposable component of the V.A.C.® Therapy system
7. Necrotic tissue with eschar present that cannot be debrided prior to subject enrollment in the study
8. Subject is exhibiting active signs and symptoms of infection of the wound(i.e. increased redness or erythema, increased pain, warmth, purulent drainage)
9. Past or current enrollment in this clinical study or any other clinical study within 30 days
10. Female Subject who is pregnant or is unwilling to use acceptable means of contraception during the duration of her participation in the study
11. Subject exhibits significant peri-wound issues that in the opinion of the investigator can interfere with the study assessments
12. Subject is unable to co-operate with study assessments or has a history of non-compliance with off-loading modalities or has a foot deformity that in the opinion of the investigator does not allow for appropriate dressing application or off loading placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - North American Center for Limb Preservation, New Haven, Connecticut
  - Drs Research Network, South Miami, Florida
  - Key Stone Medical Research Associates, Bethlehem, Pennsylvania
  - Alamo Clinical Research Consultants, San Antonio, Texas
  - Alamo Family Foot and Ankle Care, San Antonio, Texas
  - Scott and White Dept of Surgery, Temple, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- V.A.C Bridge Dressing: This is a medical device foam dressing allowing placement away from wound site. It is designed to simplify the bridging application. It is used in combination with the V.A.C. Negative Pressure Wound Therapy System. For each subject, the dressing was applied in compliance with the IFU for 48-72 hours.
Period: Overall Study
Arm/Group | V.A.C Bridge Dressing
Started | 33
Completed | 25
Not Completed | 8
Not completed — Multiple interruptions in therapy | 8

BASELINE CHARACTERISTICS:
Arm/Group | V.A.C Bridge Dressing
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White | 19
  Hispanic or Latino | 12
  American Indian or Alaskan Native | 1
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Ease of Use Assessment
Description: Each subject was assessed on the three scales (each scale was 1-Poor, 2 - Fair, 3 - Good, 4 - Excellent) and given a score on each individual characteristic (Ease of Dressing Application, Ease of Conformability, and Ease of Dressing Removal). The scores were then summed for each subject with possible range being 3-12. If the subject had a total score greater than or equal to 6, and a minimum score of greater than or equal to 2 on each individual characteristic then the subject was included in the percentage of subjects with satisfactory performance. Note that for each scale higher scores indicate better outcomes.
Time Frame: 48-72 hours (+6 hours) time period
Population: ITT (Intent to Treat) population.
Measure: Count of Participants; unit: Participants
Arm/Group | VAC GranuFoam Bridge Dressing
Number analyzed (Participants) | 30
Participants
  Ease of Dressing Application: 1-Poor | 0
  Ease of Dressing Application: 2-Fair | 3
  Ease of Dressing Application: 3-Good | 14
  Ease of Dressing Application: 4-Excellent | 13
  Ease of Comfortability: 1-Poor | 0
  Ease of Comfortability: 2-Fair | 1
  Ease of Comfortability: 3-Good | 9
  Ease of Comfortability: 4-Excellent | 20
  Ease of Dressing Removal: 1-Poor | 0
  Ease of Dressing Removal: 2-Fair | 1
  Ease of Dressing Removal: 3-Good | 4
  Ease of Dressing Removal: 4-Excellent | 25

ADVERSE EVENTS:
Time Frame: 1 week
Description: Adverse Events were assessed at each protocol scheduled visit.
Arm/Group | VAC GranuFoam Bridge Dressing
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 8/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VAC GranuFoam Bridge Dressing (N=33)
Skin Maceration (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No